CLINICAL TRIAL: NCT02562469
Title: ACTIVATE: A Computerized Training Program for Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTIVATE
Record Dates: First submitted 2015-06-03; First posted 2015-09-29 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2018-09

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACTIVATE (Experimental): ACTIVATE is a computerized neurocognitive training program (ACTIVATE; see: www.c8sciences.com) that simultaneously targets eight core neurocognitive factors (i.e., sustained attention, working memory (WM), response inhibition, speed of information processing, cognitive flexibility and control, multiple simultaneous attention, category formation, and pattern recognition and inductive thinking). ACTIVATE Is completed at home via computer with parent support. ACTIVATE intervention is conducted 3-5 times per week for between 20-30 minutes over the course or 3-4 months.
  Interventions: Other: ACTIVATE

INTERVENTIONS:
Other: ACTIVATE — A home-based computerized brain training intervention for youth.

SUMMARY:
A preliminary clinical trial of ACTIVATE will be conducted in a sample of children with ADHD. ACTIVATE is a computerized neurocognitive training program (ACTIVATE; see: www.c8sciences.com) that simultaneously targets eight core neurocognitive factors (i.e., sustained attention, working memory (WM), response inhibition, speed of information processing, cognitive flexibility and control, multiple simultaneous attention, category formation, and pattern recognition and inductive thinking).

DETAILED DESCRIPTION:
In an open clinical trial, ACTIVATE, a computer-based neurocognitive intervention will be evaluated to determine its effectiveness in improving symptoms of attention-deficit/hyperactivity disorder (ADHD) and related impairments. ACTIVATE is a computerized neurocognitive training program (ACTIVATE; see: www.c8sciences.com) that simultaneously targets eight core neurocognitive factors (i.e., sustained attention, working memory (WM), response inhibition, speed of information processing, cognitive flexibility and control, multiple simultaneous attention, category formation, and pattern recognition and inductive thinking). Youth between the ages of 7-11 will be recruited and assessed for ADHD and assigned to the ACTIVATE intervention. Assessment of outcomes will occur before, weekly during treatment, and immediately post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 7-11 with a diagnosis of ADHD
* Parent and child must be fluent English speakers
* Family has access to desktop/laptop computer at home with internet access (in order to implement the ACTIVATE intervention component, which is an online-based computer program)

Exclusion Criteria:

* Developmental delay or psychosis that impacts the child's ability to function and engage in the computerized intervention
* If the youth or parent presents with emergency psychiatric needs that require services beyond that which can be managed within a preventive intervention format (e.g. hospitalization, specialized placement outside the home)
* If the child has an estimated Full Scale IQ below 80, based on completing two subtests of the Wechsler Intelligence Scale for Children - Fourth Edition

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
ADHD symptoms on the Disruptive Behavior Rating Scale | Change in ADHD symptoms at postreatment, which is expected to occur betwen 12-18 weeks from start of treatment
  Change in ADHD symptoms over the course of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- New York University, New York, New York, United States

REFERENCES:
- See also: Families and Children Experiencing Success (FACES) Lab — http://steinhardt.nyu.edu/appsych/faceslab